CLINICAL TRIAL: NCT00863694
Title: Fecal Calprotectin in Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Steve Werlin, Professor of Pediatric Gastroenterology, M.D., Medical College of Wisconsin
Other Study IDs: calpro
Record Dates: First submitted 2009-03-16; First posted 2009-03-18 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; calprotectin; elastase
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — stool
Oversight: Data Monitoring Committee: No

SUMMARY:
Elevated fecal calprotectin is a biomarker for intestinal inflammation in cystic fibrosis

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

* Informed consent/assent not obtained

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending the cystic fibrosis clinics at the Children's Hospital of Wisconsin and Froedtert Hospital
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2009-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
collection of 150 stool specimens | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Werlin, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States